CLINICAL TRIAL: NCT02399670
Title: The Influence of Global Femoral-offset Changes After Total Hip Arthroplasty on Function, Quality of Life and Abductor Muscle Strength: a Prospective Cohort Study
Brief Title: The Influence of Global Femoral-offset Changes After Total Hip Arthroplasty
Status: Completed | Type: Observational
Sponsor: Sundsvall Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SMD_III
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Coxarthrosis
Keywords: Total hip arthroplasty; degenerative joint disease; Femoral offset; Patient reported outcome
MeSH Terms: conditions — Osteoarthritis, Hip; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Decrease femoral offset: The FO of operated side was reduced more than 5mm compared with the contralateral side.
- Restored femoral offset: The FO of operated side was within 5mm restored compared with the contralateral side.
- Increased FO: The FO of operated side was increased more than 5mm compared with the contralateral side.

SUMMARY:
The femoral-offset (FO) is one of the important perioperative parameters in THA. A prospective cohort study was conducted between September 2010 and December 2013. All patients with unilateral primary osteoarthritis (OA) treated with THA were considered for inclusion. Patients with secondary OA, previous spinal, pelvic, or lower limb injuries or fractures were excluded. Global FO was measured in each patient within 3 months before the THA and at the second postoperative day using a standardized protocol. According to the postoperative measurement, patients were divided into three groups: 1) the decreased FO group, where the FO of operated side was reduced more than 5mm compared with the contralateral side, 2) the restored FO group, where the FO of operated side was within 5mm restored compared with the contralateral side, and 3) the increased FO group, where the FO of operated side was increased more than 5mm compared with the contralateral side.

Patients were followed-up at 12 - 15 months postoperatively with self-administered WOMAC and EQ-5D questionnaires in addition to a clinical assessment with palpation of the operated hip and measurement of the abductor muscle strength.

DETAILED DESCRIPTION:
The results of total hip arthroplasty (THA) have shown great improvement during the last decades in terms of function, quality of life and prosthetic survival. Beside pain relief, surgeons aim to position the stem and cup in a correct manner to restore the biomechanical forces and range of motion of the operated hip. The femoral-offset (FO) is one of the important perioperative parameters in THA. A prospective cohort study was conducted between September 2010 and December 2013. All patients with unilateral primary osteoarthritis (OA) treated with THA were considered for inclusion. Patients with secondary OA, previous spinal, pelvic, or lower limb injuries or fractures were excluded. Global FO was measured in each patient within 3 months before the THA and at the second postoperative day using a standardized protocol. According to the postoperative measurement, patients were divided into three groups: 1) the decreased FO group, where the FO of operated side was reduced more than 5mm compared with the contralateral side, 2) the restored FO group, where the FO of operated side was within 5mm restored compared with the contralateral side, and 3) the increased FO group, where the FO of operated side was increased more than 5mm compared with the contralateral side.

Patients were followed-up at 12 - 15 months postoperatively with self-administered WOMAC and EQ-5D questionnaires in addition to a clinical assessment. Patients completed an additional questionnaire enquiring about any residual problems with the use of walking aid and residual pain around the operated hip. During the clinical assessment, palpation of the operated hip and measurement of the abductor muscle strength were undertaken.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral primary osteoarthritis treated with total hip arthroplasty

Exclusion Criteria:

* Secondary osteoarthritis
* Previous spinal, pelvic or lower limb injuries or fractures
* Bilateral osteoarthritis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with unilateral primary osteoarthritis (OA) treated with total hip arthroplasty were considered for inclusion operated between September 2010 and December 2013. Patients with secondary OA, previous spinal, pelvic, or lower limb injuries or fractures were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index | 12 months
  Patient reported functional outcome

SECONDARY OUTCOMES:
EQ-5D | 12 months
  EQ-5D that measures quality of life over 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
VAS scale | 12 months
  visual analogue scale (VAS) scale measuring pain in the operated hip during the last week-
Hip abductor muscle strength | 12 months
  and hip joint abductor muscle strength measured by electronic dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Arkan S Sayed-Noor, MD, PhD, Principal Investigator — Umeå University

REFERENCES:
- [Background] Tezuka T, Inaba Y, Kobayashi N, Ike H, Kubota S, Kawamura M, Saito T. Effects of hip joint center location and femoral offset on abductor muscle strength after total hip arthroplasty. Mod Rheumatol. 2015 Jul;25(4):630-6. doi: 10.3109/14397595.2014.988863. Epub 2014 Dec 22. PMID 25528862
- [Background] Mahmood SS, Al-Amiry B, Mukka SS, Baea S, Sayed-Noor AS. Validity, reliability and reproducibility of plain radiographic measurements after total hip arthroplasty. Skeletal Radiol. 2015 Mar;44(3):345-51. doi: 10.1007/s00256-014-2055-7. Epub 2014 Nov 18. PMID 25403426
- [Background] Berstock JR, Hughes AM, Lindh AM, Smith EJ. A radiographic comparison of femoral offset after cemented and cementless total hip arthroplasty. Hip Int. 2014 Dec 5;24(6):582-6. doi: 10.5301/hipint.5000160. Epub 2014 Sep 1. PMID 25198306
- [Background] Sariali E, Klouche S, Mouttet A, Pascal-Moussellard H. The effect of femoral offset modification on gait after total hip arthroplasty. Acta Orthop. 2014 Apr;85(2):123-7. doi: 10.3109/17453674.2014.889980. Epub 2014 Feb 25. PMID 24564749
- [Background] Hayashi S, Nishiyama T, Fujishiro T, Hashimoto S, Kanzaki N, Nishida K, Kuroda R, Kurosaka M. Excessive femoral offset does not affect the range of motion after total hip arthroplasty. Int Orthop. 2013 Jul;37(7):1233-7. doi: 10.1007/s00264-013-1881-x. Epub 2013 Apr 5. PMID 23553118
- [Background] Chamnongkich S, Asayama I, Kinsey TL, Mahoney OM, Simpson KJ. Difference in hip prosthesis femoral offset affects hip abductor strength and gait characteristics during obstacle crossing. Orthop Clin North Am. 2012 Nov;43(5):e48-58. doi: 10.1016/j.ocl.2012.07.008. Epub 2012 Sep 15. PMID 23102422
- [Background] Cassidy KA, Noticewala MS, Macaulay W, Lee JH, Geller JA. Effect of femoral offset on pain and function after total hip arthroplasty. J Arthroplasty. 2012 Dec;27(10):1863-9. doi: 10.1016/j.arth.2012.05.001. Epub 2012 Jul 17. PMID 22810007
- [Result] Mahmood SS, Mukka SS, Crnalic S, Wretenberg P, Sayed-Noor AS. Association between changes in global femoral offset after total hip arthroplasty and function, quality of life, and abductor muscle strength. A prospective cohort study of 222 patients. Acta Orthop. 2016 Feb;87(1):36-41. doi: 10.3109/17453674.2015.1091955. Epub 2015 Oct 16. PMID 26471772